CLINICAL TRIAL: NCT06737627
Title: Development and Validation of the Observatory Battery of Common Eye Disorders for Adults With Intellectual Disability
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202212036RINA
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Intellectual Disability
Keywords: Intellectual disability, Adults, Visual Scale, Caregiver
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intellectual disability
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Background:

Around 15% of the global population has some form of disability. Rights to obtain proper health care is an emphasis in the United Nationals Convention on the Right of People with Disability. Due to the importance of improving vision health for people with disabilities, studies on how to identify vision problems becomes extremely important in policy formulation for all countries. Among all types of disabilities, people with intellectual disability (ID) are among the ones where vision problems are the hardest to detect.

Currently, no caregiver assessable scales are available, as a result, adults with ID are at high risk of delayed diagnose for common ocular conditions. Objectives: This is a one-year project.

The objective of this study is two folds:

1. To develop an item bank of ocular conditions of adults with ID;
2. To develop a scale for caregivers to detect ocular conditions for adults with ID, and to validate the reliability, construct validity and responsiveness of the scale.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 and above
2. Primary caregivers for at least one adult with ID (have disability identification or (and) certification).

Exclusion Criteria:

1. Unable to communicate in Mandarin or Taiwanese.(Primarycaregivers)
2. Unable to cooperate with eye examination.(ID)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Intellectual disability
Sampling Method: Non-Probability Sample
Enrollment: 740 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2026-01-29 (Estimated)

PRIMARY OUTCOMES:
Collection of Socioeconomic Data for Individuals with Disabilities | 1-3 months
  This study collects basic socioeconomic data of individuals with disabilities through tailored questionnaires, including gender, date of birth, educational background, living conditions, and employment status. The questionnaire is designed to accommodate the specific characteristics of individuals with intellectual disabilities and is completed by respondents or their proxies. These data will be analyzed to understand the impact of socioeconomic factors on the visual health and accessibility to medical services for people with disabilities. Ethical guidelines are strictly followed to ensure confidentiality and protect participant rights.
Assessment Scales for Individuals with Disabilities | 1-3 months
  This study utilizes validated assessment tools to evaluate the visual functions and daily living abilities of individuals with disabilities. These include the Activities of Daily Living (ADL) Scale and Instrumental Activities of Daily Living (IADL) Scale, supplemented by specific observational items for visual health and related functional behaviors. The scales employ a graded scoring system covering personal hygiene, mobility, social interaction, and visual challenges. The collected data will help analyze the impact of visual impairment on independent living skills and support the development of tailored visual intervention strategies. Participant privacy and ethical compliance are rigorously maintained.
Ophthalmologic Examination Form | 1-3 months
  A standardized ophthalmologic examination form is employed in this study to record detailed visual and eye health data of individuals with disabilities. The form includes uncorrected and corrected visual acuity, intraocular pressure, eye movement, corneal conditions, iris, macula, retina, and other ocular components. It also documents spherical power, cylindrical power, and axis to assess refractive correction needs. The form provides a section for medical recommendations such as eyeglass prescription, medical referral, or regular follow-up. These comprehensive data support analysis of visual problems' effects on individuals and guide the formulation of personalized visual intervention plans.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Care facility, New Taipei City
  - Care facility, Taipei